CLINICAL TRIAL: NCT00667745
Title: Lithium Use for Bipolar Disorder (LiTMUS): A Randomized Controlled Effectiveness Trial
Brief Title: Effectiveness of Lithium Plus Optimized Medication in Treating People With Bipolar Disorder
Acronym: LiTMUS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N01 MH080001-01; DSIR AT; N01MH080001 (NIH)
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Results first posted 2013-06-28 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2010-07

CONDITIONS: Bipolar Disorder
Keywords: Lithium; Symptoms; Medication Changes
MeSH Terms: conditions — Bipolar Disorder | interventions — Lithium Carbonate; Lithium

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants received lithium plus optimized medication treatment, as needed.
  Interventions: Drug: Lithium Carbonate; Drug: Optimized Treatment (OPT)
- 2 (Active Comparator): Participants only received optimized medication treatment, as needed; lithium was not be used.
  Interventions: Drug: Optimized Treatment (OPT)

INTERVENTIONS:
Drug: Lithium Carbonate — Lithium was started at 300 mg and then increased to 600 mg after 3 days. Lithium doses were maintained at 600 mg per day for 8 weeks, but may have been adjusted after that time as needed up to a serum level of 1.2 mEq/L.
  Other Names: Lithium
  Arms: 1
Drug: Optimized Treatment (OPT) — The foundation of OPT was to maintain treatment that will typically include at least one FDA-approved mood stabilizer other than lithium (e.g., divalproex, carbamazepine, risperidone, quetiapine, olanzapine, aripiprazole, ziprasidone) and to follow the recommendations summarized in the evidence-based stages of the Texas Implementation of Medication Algorithm (TIMA) revised guidelines.

SUMMARY:
This study evaluated whether lithium included as part of optimized medication treatment improved overall level of illness, symptoms of mania and depression, and quality of life in people with bipolar disorder.

DETAILED DESCRIPTION:
Bipolar illness, a brain disorder that causes dramatic changes in a person's mood and energy, affects about 2.6% of adults in the United States. Bipolar disorder is characterized by cyclical periods of extreme highs and lows, known as episodes of mania and depression. A person undergoing an episode of mania often experiences euphoric moods, increased energy, and aggressive behaviors, while a person in a depressed state often experiences low moods, lack of energy, and feelings of sadness. Lithium is a widely used mood stabilizing medication that has been shown to reduce the occurrence and intensity of manic episodes and may lessen depressive episodes as well. Including lithium as a part of a personalized medication treatment approach may be the most effective means of improving symptoms of bipolar disorder. This study will evaluate whether lithium included as part of optimized medication treatment improves overall level of illness, symptoms of mania and depression, and quality of life in people with bipolar disorder.

Participation in this study lasted for 6 months. All participants had an initial assessment that included an interview and questionnaires to confirm a diagnosis of bipolar disorder, vital sign measurements, a blood draw, and if female, pregnancy. Eligible participants were then assigned randomly to receive either optimized medication plus lithium or optimized medication without lithium. Participants in both groups received 6 months of monitored treatment with their medication regimens, as prescribed by their study doctor. Participants attended study visits every 2 weeks for the first 8 weeks and then once a month for 4 more months. These visits lasted between 45 and 60 minutes and included medication adjustments and questions about symptoms, side effects, and quality of life.

We would like to acknowledge that medication was kindly donated by Ortho-McNeil Janssen Scientific Affairs, LLC.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV Criteria for bipolar disorder (type I or II)
* Currently symptomatic, as defined as a Clinical Global Impressions Scale-Bipolar Version, Overall Severity Index (CGI-BP-S) of greater than or equal to 3
* If taking or has taken lithium, must be off lithium for at least 30 days before study entry
* If a woman of child bearing potential, agrees to inform their doctor at the earliest possible time of their plans to conceive, to use adequate contraception (e.g. oral contraceptives, intrauterine device, barrier methods, total abstinence from intercourse), and to acknowledge the risks of lithium to the fetus and infant (Depo Provera is acceptable if it is started 3 months before study entry)

Exclusion Criteria:

* Renal impairment (serum creatinine greater than 1.5 mg/dL)
* Thyroid stimulating hormone (TSH) over 20% above the upper normal limit (participants maintained on thyroid medication must be euthyroid for at least 3 months before Visit 1)
* History of lithium toxicity that was not caused by mismanagement or overdose
* Other contraindication to lithium (e.g., hypersensitivity to lithium or any component of the formulation, severe cardiovascular or renal disease, severe debilitation, dehydration, sodium depletion, pregnancy)
* Currently in crisis such that inpatient hospitalization or other crisis - Participated in a clinical trial of an investigational drug within the 1 months before study entry
* Pregnant or breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Start 2008-04; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Stanford University, Stanford, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Case Western Reserve University, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Texas Health Science Center, San Antonio, Texas

REFERENCES:
- [Derived] Ostacher MJ, Nierenberg AA, Rabideau D, Reilly-Harrington NA, Sylvia LG, Gold AK, Shesler LW, Ketter TA, Bowden CL, Calabrese JR, Friedman ES, Iosifescu DV, Thase ME, Leon AC, Trivedi MH. A clinical measure of suicidal ideation, suicidal behavior, and associated symptoms in bipolar disorder: Psychometric properties of the Concise Health Risk Tracking Self-Report (CHRT-SR). J Psychiatr Res. 2015 Dec;71:126-33. doi: 10.1016/j.jpsychires.2015.10.004. Epub 2015 Oct 9. PMID 26476489
- [Derived] Reilly-Harrington NA, Sylvia LG, Leon AC, Shesler LW, Ketter TA, Bowden CL, Calabrese JR, Friedman ES, Ostacher MJ, Iosifescu DV, Rabideau DJ, Thase ME, Nierenberg AA. The Medication Recommendation Tracking Form: a novel tool for tracking changes in prescribed medication, clinical decision making, and use in comparative effectiveness research. J Psychiatr Res. 2013 Nov;47(11):1686-93. doi: 10.1016/j.jpsychires.2013.07.009. Epub 2013 Jul 30. PMID 23911057
- [Derived] Beech RD, Leffert JJ, Lin A, Sylvia LG, Umlauf S, Mane S, Zhao H, Bowden C, Calabrese JR, Friedman ES, Ketter TA, Iosifescu DV, Reilly-Harrington NA, Ostacher M, Thase ME, Nierenberg A. Gene-expression differences in peripheral blood between lithium responders and non-responders in the Lithium Treatment-Moderate dose Use Study (LiTMUS). Pharmacogenomics J. 2014 Apr;14(2):182-91. doi: 10.1038/tpj.2013.16. Epub 2013 May 14. PMID 23670706
- [Derived] Nierenberg AA, Friedman ES, Bowden CL, Sylvia LG, Thase ME, Ketter T, Ostacher MJ, Leon AC, Reilly-Harrington N, Iosifescu DV, Pencina M, Severe JB, Calabrese JR. Lithium treatment moderate-dose use study (LiTMUS) for bipolar disorder: a randomized comparative effectiveness trial of optimized personalized treatment with and without lithium. Am J Psychiatry. 2013 Jan;170(1):102-10. doi: 10.1176/appi.ajp.2012.12060751. PMID 23288387
- [Derived] Sylvia LG, Reilly-Harrington NA, Leon AC, Kansky CI, Ketter TA, Calabrese JR, Thase ME, Bowden CL, Friedman ES, Ostacher MJ, Iosifescu DV, Severe J, Keyes M, Nierenberg AA. Methods to limit attrition in longitudinal comparative effectiveness trials: lessons from the Lithium Treatment - Moderate dose Use Study (LiTMUS) for bipolar disorder. Clin Trials. 2012 Feb;9(1):94-101. doi: 10.1177/1740774511427324. Epub 2011 Nov 10. PMID 22076437

RESULTS

PARTICIPANT FLOW:
Groups:
- OPT With Lithium: Participants received lithium plus optimized medication treatment, as needed.
  Lithium Carbonate : Lithium was started at 300 mg and then increased to 600 mg after 3 days. Lithium doses were maintained at 600 mg per day for 8 weeks, but may have been adjusted after that time as needed up to a serum level of 1.2 mEq/L.
  Optimized Treatment (OPT) : The foundation of OPT was to maintain treatment that will typically include at least one FDA-approved mood stabilizer other than lithium (e.g., divalproex, carbamazepine, risperidone, quetiapine, olanzapine, aripiprazole, ziprasidone) and to follow the recommendations summarized in the evidence-based stages of the Texas Implementation of Medication Algorithm (TIMA) revised guidelines.
- OPT Without Lithium: Participants only received optimized medication treatment, as needed; lithium was not be used.
  Optimized Treatment (OPT) : The foundation of OPT was to maintain treatment that will typically include at least one FDA-approved mood stabilizer other than lithium (e.g., divalproex, carbamazepine, risperidone, quetiapine, olanzapine, aripiprazole, ziprasidone) and to follow the recommendations summarized in the evidence-based stages of the Texas Implementation of Medication Algorithm (TIMA) revised guidelines.
Period: Overall Study
Arm/Group | OPT With Lithium | OPT Without Lithium
Started | 141 | 142
Completed | 116 | 121
Not Completed | 25 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OPT With Lithium | OPT Without Lithium | Total
Number analyzed (Participants) | 141 | 142 | 283
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 141 | 142 | 283
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.7 (11.7) | 39.4 (13.0) | 39.1 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 83 | 160
  Male | 64 | 59 | 123
Region of Enrollment [Number; unit: participants]
  United States | 141 | 142 | 283

OUTCOME MEASURES:

1. Primary Outcome: Overall Change in Bipolar Illness Severity as Measured by Clinical Global Impression for Bipolar Disorder Severity (CGI-BP-S) Score
Description: Scale: Clinical Global Impression for Bipolar Disorder Severity (CGI-BP-S) Construct: This scale holistically measures severity of a participant's depression, mania, and overall illness.
  Range: 0- not assessed, 1-normal (not at all ill), 2- borderline mentally ill, 3- mildly ill, 4- moderately ill, 5- markedly ill, 6- severely ill, 7- among the most extremely ill patients.
Time Frame: Relevant time points: baseline and week 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OPT With Lithium | OPT Without Lithium
Number analyzed (Participants) | 141 | 142
units on a scale | -1.22 (1.50) | -1.48 (1.37)
Statistical Analysis 1: Comparison: OPT With Lithium vs OPT Without Lithium; Test type: Superiority; p = 0.33, Mixed Models Analysis; F value, main effect = 0.94

2. Primary Outcome: Number of Necessary Medication Adjustments
Description: Metric Definition (Necessary Clinical Adjustments (NCA)): Medication adjustments to reduce symptoms, optimize treatment response and functioning, or to address intolerable side effects. This was determined with the Medication Recommendation Tracking Form (MRTF), a novel method for capturing physician prescribing behavior and clinical decision making.
  Range: whole numbers
  Relevant time points: Weeks 2, 4, 6, 8, 12, 16, 20, and 24.
Time Frame: Measured over 6 months
Measure: Mean (Standard Deviation); unit: Adjustments
Arm/Group | OPT With Lithium | OPT Without Lithium
Number analyzed (Participants) | 141 | 142
Adjustments | 1.17 (0.96) | 1.26 (1.11)
Statistical Analysis 1: Comparison: OPT With Lithium vs OPT Without Lithium; Test type: Superiority; p = 0.967, Chi-squared; Chi-squared = 0.00

3. Secondary Outcome: Depression Symptoms as Measured Self Report Montgomery Asberg Depression Rating Scale (MADRS)
Description: The MADRS is a 10-item measure and has a fixed scaling of seven points (from 0 through 6), with 0 representing sypmtoms that are not present and 6 being the most severe symptoms. When completed, the sum of each individual item is taken to create an overall score.
  Overall scores:
  0 to 6 - normal /symptom absent 7 to 19 - mild depression 20 to 34 - moderate depression >34 - severe depression
Time Frame: Measured over 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OPT With Lithium | OPT Without Lithium
Number analyzed (Participants) | 141 | 142
units on a scale | 8.20 (12.29) | 8.84 (13.59)
Statistical Analysis 1: Comparison: OPT With Lithium vs OPT Without Lithium; Test type: Superiority; p = 0.50, Mixed Models Analysis; Mean Difference (Net) = 0.45

4. Secondary Outcome: Mania Symptoms as Measured by the Young Mania Rating Scale (YMRS)
Description: The scale has 11 items and is based on the patient's subjective report of his or her clinical condition over the previous 48 hours. There are four items that are graded on a 0 to 8 scale with 0 indicating that symptoms are absent and 8 indicating that symptoms are severe (irritability, speech, thought content, and disruptive/aggressive behavior), while the remaining seven items are graded on a 0 to 4 scale, with 0 indicating that symptoms are absent and 4 indicating that symptoms are severe (Elevated mood, increased motor activity-energy, sexual interest, sleep, language-thought disorder, appearance, and insight). Total scores can vary from 0-60, with 0 indicating that symptoms are completely absent and 60 indicating that the patient is severely manic.
Time Frame: Measured over 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OPT With Lithium | OPT Without Lithium
Number analyzed (Participants) | 141 | 142
units on a scale | 6.35 (10.09) | 5.79 (8.45)
Statistical Analysis 1: Comparison: OPT With Lithium vs OPT Without Lithium; Test type: Superiority; p = 0.88, Mixed Models Analysis; Mean Difference (Net) = 0.02

5. Secondary Outcome: Suicidality as Measured by the Modified Scale for Suicidal Ideation (MSSI)
Description: The Modified Scale for Suicide Ideation (MSSI) assesses the presence of absence of suicide ideation and the degree of severity of suicidal ideas. The time frame is from the point of interview and the previous 48 hours. It uses 13 items from the Scale for Suicidal Ideation (SSI) and 5 new items. The modifications increased both reliability and validity. The scale was also changed to range from 0 to 3, yielding a total score ranging from 0 to 54. A total score is attained by summing all of the items. A score between 0-8 indicates low suicidal ideation; 9-20 indiciates mild-moderate suicidal ideation; 21+ indicates severe suicidal ideation.
Time Frame: Measured over 6 months
Measure: Mean (Standard Deviation); unit: units of scale
Arm/Group | OPT With Lithium | OPT Without Lithium
Number analyzed (Participants) | 141 | 142
units of scale | 0.73 (4.12) | 1.10 (3.77)
Statistical Analysis 1: Comparison: OPT With Lithium vs OPT Without Lithium; Test type: Superiority; p = .49, Mixed Models Analysis — Value shown above describes emergent suicidal ideation for participants with baseline MSSI = 0. P=.36 describes exacerbation of baseline suicidal ideation for those with baseline MSSI > 0; Mean Difference (Net) = .92

ADVERSE EVENTS:
Arm/Group | OPT With Lithium | OPT Without Lithium
Serious Adverse Events (participants affected / at risk) | 14/141 | 12/142
Other Adverse Events (participants affected / at risk) | 69/141 | 61/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OPT With Lithium (N=141) | OPT Without Lithium (N=142)
Alcohol Detoxification (Psychiatric disorders) | 1 (1) | 0 (0)
Cholecystitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Chron's Disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dehydration (General disorders) | 1 (1) | 0 (0)
Mania (Psychiatric disorders) | 2 (2) | 2 (2)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumonia (Nervous system disorders) | 1 (1) | 0 (0)
Pregnancy (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 4 (4) | 6 (6)
Breast Cancer (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Fluid Retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Upper limb fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OPT With Lithium (N=141) | OPT Without Lithium (N=142)
Aches/pains (Musculoskeletal and connective tissue disorders) | 13 (15) | 8 (9)
Diarrhea/gastrointestinal distress (Gastrointestinal disorders) | 14 (21) | 5 (6)
Fatigue/sedation/drowsiness (General disorders) | 20 (20) | 19 (25)
Dizziness/Headaches (General disorders) | 8 (9) | 13 (19)
Memory/Concentration/Cognitive Impairment (Psychiatric disorders) | 10 (11) | 1 (1)
Tremors (Musculoskeletal and connective tissue disorders) | 14 (14) | 7 (7)
Increased appetite/weight gain (Metabolism and nutrition disorders) | 15 (15) | 15 (16)
Dry mouth/thirst (General disorders) | 8 (8) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No